CLINICAL TRIAL: NCT03117621
Title: An Observational Study of Blinatumomab Safety and Effectiveness, Utilization, and Treatment Practices
Brief Title: Observational Study of Blinatumomab
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20150136
Record Dates: First submitted 2017-03-06; First posted 2017-04-18 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Blincyto Use in Routine Clinical Practice
Keywords: Blincyto

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients initiating Blinatumomab: Patients initiating Blinatumomab after Country-Specific Reimbursement approval in routine clinical practice.

SUMMARY:
An observational study of blinatumomab safety and effectiveness, utilisation, and treatment practices.

DETAILED DESCRIPTION:
The primary objective of this study is to characterize the safety of Blincyto in routine clinical practice. Blincyto effectiveness, medication errors, and utilisation; and select healthcare resource use while using Blincyto will also be described. Safety and effectiveness of Blincyto in specified subgroups of patients will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

- Medical records of patients initiating Blincyto after country-specific reimbursement in routine clinical practice will be eligible for extraction.

Exclusion Criteria:

* Medical records of patients who have participated in Blincyto clinical trials will be excluded since their treatment will be prescribed by the study protocol unless the patient is receiving new Blincyto treatment outside the clinical trial.
* Medical records of patients participating in other Amgen non-interventional prospective studies in which safety endpoints are collected will be excluded.
* Medical records of patients who have received Blincyto via an expanded access/compassionate use program will be excluded.
* In countries where patient informed consent is required for access to their medical records, any patient who does not provide informed consent will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include patients receiving Blincyto at participating clinical centres after country-specific reimbursement of Blincyto in the Europe.
Sampling Method: Non-Probability Sample
Enrollment: 279 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with specified AEs as mentioned in description | Estimated to be 100 days
  * Neurological adverse events
  * Opportunistic infections
  * Cytokine release syndrome
Time to onset of first specified AEs | Estimated to be 100 days
  Time to onset of first specified AEs.
Summary of duration of specified AEs as detailed in the description (all events and resolved/recovered events) | Estimated to be 100 days
  Summary of duration of specified AEs (all events and resolved/recovered events)
  * Neurological adverse events
  * Opportunistic Infections
Proportion of Blincyto administrations with medication errors | Estimated to be 100 days
  Proportion of Blincyto administrations with medication errors, defined as an unintended failure in the drug treatment process that leads to, or has the potential to lead to, harm to the patient, identified through medical records. Types of medication errors will also be described
  * incorrect Blincyto dose administered/prepared (eg. drug concentration, device issues, treatment according to SmPC)
  * does not include treatment related to dexamethasone.

SECONDARY OUTCOMES:
Proportion of patients with AEs as detailed in the description | Estimated to be 100 days
  Incidence of all AEs collected in this study (overall, and by severity and seriousness) occurring during blinatumomab treatment and up to 30 days after completion of treatment
  • Incidence of specified AEs and all AEs collected in this study among patient subgroups defined by demographic and clinical factors.
Proportion of patients achieving Complete Remission overall and amongst patient sub-groups | Estimated to be 100 days
  * Proportion of patients achieving Complete Remission within 2 cycles of Blincyto treatment
  * Complete remission - Defined as ≤ 5% bone marrow myeloblasts, platelets more than 100,000 cells per µL, and absolute neutrophil count > 1,000 cells per µL.
Proportion of patients achieving CR/CRh*/CRi amongst patient sub-groups | Estimated to be 100 days
  Proportion of patients achieving CR/CRh*/CRi within 2 cycles Blincyto treatment
  * CR defined as ≤ 5% bone marrow blasts, platelets more than 100,000 cells per µL, and absolute neutrophil count > 1,000 cells per µL
  * CRh* defined as ≤ 5% bone marrow blasts, platelets more than 50,000 cells per µL, and absolute neutrophil count > 500 cells per µL
  * CRi defined as ≤ 5% bone marrow blasts and incomplete recovery of peripheral blood counts.
Proportion of patients receiving allogeneic HSCT amongst patient sub-groups | Estimated to be 100 days
  Proportion of patients receiving allogeneic HSCT amongst patient sub-groups. Defined for the subset of subjects who achieved CR.
1-year and 100-day mortality proportion after allogeneic HSCT amongst patient sub-groups | Estimated to be 100 days
  1-year and 100-day mortality proportion after allogeneic HSCT amongst patient sub-groups. Defined for the subset of subjects who achieved CR.
Relapse-free survival (RFS) time amongst patient sub-groups | Estimated to be 100 days
  Relapse-free survival (RFS) time - defined as time from CR/CRh*/CRi until relapse (proportion of blasts in bone marrow > 5% or blasts in peripheral blood after documented CR/CRh*/CRi) or death. Defined for the subset of subjects who achieved CR.
Disease Free Survival (DFS) time | Estimated to be 100 days
  Disease Free Survival time - Defined as time from initiation of Blincyto (for MRD positive patients at initiation) until date of relapse or death.
Overall survival (OS) time amongst patient sub-groups | Estimated to be 100 days
  Overall survival (OS) time - defined as time from initiation of Blincyto until death.
Proportion of patients with MRD achieving CR/CRh*/CRi within 2 cycles of Blincyto | Estimated to be 100 days
  Overall and amongst patient sub-groups - Proportion of patients with minimal residual disease (MRD) among those who achieve CR/CRh*/CRi within two cycles of Blincyto treatment - hematologic MRD detected by polymerase chain reaction (PCR) (or flow cytometry) at a level of
  1 x 10-4 or higher.
Blincyto utilisation: Number of completed cycles | Estimated to be 100 days
Blincyto utilisation: Total number of days of administration | Estimated to be 100 days
Blincyto utilisation: Proportion of patients with dose step-up on Day 8 | Day 8
Blincyto utilisation: Number of cycles initiated | Estimated to be 100 days
Blincyto utilisation: Number of bag changes | Estimated to be 100 days
Blincyto utilisation: Proportion of patients with treatment changes | Estimated to be 100 days
  Treatment changes include interruption, discontinuation, and dose reduction.
Select healthcare resource use: Number of bag changes in each setting | Estimated to be 100 days
  Setting of blincyto bag changes include in the hospital, in the outpatient clinic, or at home.
Select healthcare resource use: Total number of days of inpatient Blincyto treatment | Estimated to be 100 days
Select healthcare resource use: Proportion of treatment days that were inpatient | Estimated to be 100 days
Select healthcare resource use: Incidence of hospitalization not related to infusion | Estimated to be 100 days
Select healthcare resource use: Length of hospital stay not related to infusion | Estimated to be 100 days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (80):
- Austria (3):
  - Ordensklinikum Linz Elisabethinen, Linz
  - Landeskrankenhaus Salzburg, Salzburg
  - Hanuschkrankenhaus, Vienna
- Czechia (3):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Plzen, Pilsen
  - Ustav hematologie a krevni transfuze, Prague
- Helsinki University Central Hospital, Helsinki, Finland
- France (15):
  - Centre Hospitalier Universitaire Dieu Angers, Angers
  - Centre Hospitalier Regional Universitaire de Besancon, Hopital Jean Minjoz, Besançon
  - Hopital d Instruction des Armee, Clamart
  - Centre Hospitalier Universitaire de Clermont Ferrand - Hopital Estaing, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - Centre Hospitalier Régional Universitaire de Lille - Hôpital Claude Huriez, Lille
  - Centre Hospitalier Universitaire de Montpellier - Hopital Saint Eloi, Montpellier
  - Centre Hospitalier Universitaire de Nice, Nice
  - Hopital Saint Louis, Paris
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Haut Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Poitiers - Hopital la Miletrie, Poitiers
  - Institut de Cancerologie Strasbourg, Strasbourg
  - Centre Hospitalier Universitaire de Toulouse - Hopital Purpan, Toulouse
  - Centre Hospitalier Universitaire de Nancy - Hopital de Brabois, Vandœuvre-lès-Nancy
- Germany (5):
  - Universitätsklinikum Dresden, Dresden
  - Klinikum und Fachbereich Medizin Johann Wolfgang Goethe-Universität Frankfurt am Main, Frankfurt am Main
  - Universitätsklinikum Halle/Saale, Halle
  - Städtisches Klinikum München GmbH, München
  - Klinikum Oldenburg AoR, Oldenburg
- Greece (4):
  - Evangelismos Hospital, Athens
  - Laiko General Hospital of Athens, Athens
  - Attikon University Hospital, Athens
  - University Hospital of Patras, Pátrai
- Italy (19):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliera Universitaria di Bologna Policlinico S Orsola Malpighi, Bologna
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera Universitaria Policlinico Vittorio Emanuele Presidio Ospedaliero G Rodolico, Catania
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Ospedale Policlinico San Martino IRCCS, Genova
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliero Universitaria di Modena, Modena
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Presidio Ospedaliero Andrea Tortora, Pagani (SA)
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera di Perugia Ospedale Santa Maria della Misericordia, Perugia
  - Azienda Unita Sanitaria Locale Pescara Ospedale Civile Santo Spirito, Pescara
  - Azienda Unita Sanitaria Locale Istituto di Ricovero di Reggio Emilia Arcispedale Santa Maria Nuova, Reggio Emilia
  - Azienda Ospedaliera Policlinico Umberto I, Roma
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino Ospedale Molinette, Torino
  - Azienda Ospedaliera Ordine Mauriziano - Presidio Umberto I, Torino
  - Azienda Unità Locale Socio Sanitaria 3 Ospedale Dell Angelo, Venezia
- Netherlands (3):
  - Academisch Medisch Centrum, Amsterdam
  - Erasmus Medical Center, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (6):
  - SPZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - Szpital Specjalistyczny imienia Ludwika Rydygiera w Krakowie Sp zoo, Krakow
  - Szpital Kliniczny im H Swiecickiego Uniwersytetu Medycznego im K Marcinkowskiego w Poznaniu, Poznan
  - Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu Medycznego, Warsaw
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - Uniwersytecki Szpital Kliniczny im Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw
- Portugal (4):
  - Instituto Portugues de Oncologia de Lisboa Francisco Gentil, EPE, Lisbon
  - Centro Hospitalar de Lisboa Central, EPE - Hospital de Santo Antonio dos Capuchos, Lisbon
  - Centro Hospitalar Universitário de Lisboa Norte, EPE - Hospital Santa Maria, Lisbon
  - Centro Hospitalar do Porto EPE - Hospital de Santo Antonio, Porto
- Akademiska Sjukhuset, Uppsala, Sweden
- Switzerland (9):
  - Kantonsspital Aarau, Aarau
  - Universitaetsspital Basel, Basel
  - Instituto Oncologico Della Svizzera Italiana, Bellinzona
  - Inselspital Bern, Bern
  - Hopitaux Universitaires de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital St Gallen, Sankt Gallen
  - Universitaetsspital Zuerich, Zurich
- United Kingdom (7):
  - Northwick Park Hospital, Harrow
  - St James University Hospital, St James Institute of Oncology, Leeds
  - Royal Liverpool University Hospital, Liverpool
  - St Bartholomews Hospital, London
  - St Georges Hospital, London
  - Manchester Royal Infirmary, Manchester
  - Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com